CLINICAL TRIAL: NCT00238277
Title: Phase II Study of Temozolomide and Radiation in Newly Diagnosed GBM Patients After Resection and Insertion of Gliadel® Wafers
Brief Title: Temozolomide During and After Radiation Therapy in Treating Patients Who Have Undergone Previous Surgery and Placement of Gliadel Wafers for Newly Diagnosed Glioblastoma Multiforme
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated - due to low accrual
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: J0498; P30CA006973 (NIH); CDR0000445270; 04-12-16-03 (Other: JHM IRB)
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Temozolomide; Chemotherapy, Adjuvant; Drug Therapy; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: temozolomide
Procedure: adjuvant therapy
Procedure: chemotherapy
Procedure: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving temozolomide during and after radiation therapy may kill any tumor cells that remain after surgery and placement of Gliadel wafers.

PURPOSE: This phase II trial is studying how well giving temozolomide during and after radiation therapy works in treating patients who have undergone previous surgery and placement of Gliadel wafers for newly diagnosed glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of adjuvant temozolomide when administered during and after external beam radiotherapy, in terms of survival, in patients with newly diagnosed glioblastoma multiforme who have undergone prior total surgical resection and placement of polifeprosan 20 with carmustine implant (Gliadel® wafers).

OUTLINE: This is an open-label study.

Patients undergo external beam radiotherapy 5 days a week for 6 weeks and concurrently receive oral temozolomide once daily for 6 weeks. No more than 28 days later, patients receive additional oral temozolomide once daily on days 1-5. Treatment with temozolomide repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 2 months for survival.

PROJECTED ACCRUAL: A total of 72 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed supratentorial grade IV astrocytoma (glioblastoma multiforme)
* Underwent gross total resection within the past 6 weeks

  * Postoperative contrast-enhancing tumor extends ≤ 1 cm from the margin of the surgical cavity
  * 6-8 polifeprosan 20 with carmustine implants (Gliadel® wafers) were placed in the surgical resection cavity at time of surgery

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 mg/dL
* Transaminases ≤ 4 times upper limit of normal

Renal

* Creatinine ≤ 1.7 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known hypersensitivity reaction to temozolomide
* No other malignancy within the past 5 years except curatively treated carcinoma in situ or basal cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior immunotherapy for the brain tumor
* No prior biologic agents (e.g., immunotoxins, immunoconjugates, antisense agents, peptide-receptor agonists, interferons, interleukins, tumor-infiltrating lymphocyte therapy, lymphokine-activated killer cell therapy, or gene therapy) for the brain tumor

Chemotherapy

* See Disease Characteristics
* No other prior chemotherapy for the brain tumor

Endocrine therapy

* No prior hormonal therapy for the brain tumor
* Prior glucocorticoid therapy allowed

Radiotherapy

* No prior radiotherapy for the brain tumor

Surgery

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-02-15 (Actual); Primary Completion 2007-12-11 (Actual); Study Completion 2007-12-11 (Actual)

PRIMARY OUTCOMES:
Death

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A. Grossman, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States